CLINICAL TRIAL: NCT03250403
Title: Efficacy of Platelet Rich Plasma Injection in Diabetic Neuropathy: Double Blinded Randomized Controlled Trial
Brief Title: Efficacy of Platelet Rich Plasma Injection in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Prenciple investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: peripheral neuropathy PRP
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP injection (Experimental)
  Interventions: Drug: PRP injection; Other: traditional medical treatment
- medical treatment (Active Comparator)
  Interventions: Other: traditional medical treatment

INTERVENTIONS:
Drug: PRP injection — peri-neural injection of platelet rich plasma
  Arms: PRP injection
Other: traditional medical treatment — traditional medical treatment

SUMMARY:
To evaluate the clinical efficacy and safety of peri-neural platelet rich plasma (PRP) injection in the treatment of diabetic peripheral neuropathy compared to traditional medical treatment.

DETAILED DESCRIPTION:
Background: Neuropathy is a common complication of diabetes mellitus (DM) with a wide clinical spectrum that encompasses generalized to focal and multifocal forms not only leads to an impaired quality of life, but also to an increased morbidity and mortality . Till now there is no available effective therapy for the treatment of diabetic peripheral neuropathy (DPN). Autologous platelet-rich plasma is easy and cost-effective method as it provides necessary growth factors that promote wound healing/growth, angiogenesis, and axon regeneration .

Objective: To evaluate the clinical efficacy and safety of peri-neural platelet rich plasma (PRP) injection in the treatment of diabetic peripheral neuropathy compared to traditional medical treatment.

Method : Prospective double blinded randomized controlled trial was conducted . All included patients had type 2 DM selected from Endocrinology unit Department of Internal medicine, Assuit university Hospital, Egypt . DPN of at least 5 years duration of symptoms . Patients with other causes of neuropathy like hereditary neuropathies , entrapment neuropathies ,connective tissue diseases , vertebral diseases ,thyroid disorders and end organ failure were excluded . Neuropathy was assessed by the modified Toronto Clinical Neuropathy Score (mTCNS) 2001 (3) , Baseline pain and nerve conduction studies were done. Then they were double blindly divided into two groups, Group I underwent PRP preineural injection under ultrasound guidance plus medical treatment . Group װreceived medical treatment only( control group) . Blood glucose was strictly controlled in both groups . Patients were followed every month for 3 months by mTCNS and by nerve conduction studies. Results were expressed as means ± standard deviation or frequencies. Independent Student's t test was done for comparison between groups

ELIGIBILITY:
Inclusion Criteria:

* Diabetic peripheral neuropathy of at least 5 years duration of symptoms

Exclusion Criteria:

* hereditary neuropathies , entrapment neuropathies , connective tissue diseases , vertebral diseases , thyroid disorders and end organ failure

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Numbness | 6 months
  modified Toronto Clinical Neuropathy Score
pain | 6 months
  VAS 0-10 scale

SECONDARY OUTCOMES:
Conduction velocity | 6 months
  Meter/second

CONTACTS AND LOCATIONS:
Overall Officials: Abdelraheem M Alawaamy, Dr, Principal Investigator — Assiut University
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided